CLINICAL TRIAL: NCT06780345
Title: Role of Vitamin C Infusion in Postoperative Mechanically Ventilated Neonates With Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amany Mohamed Abotaleb, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR117/2/23
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Vitamin C; Postoperative; Mechanically Ventilation; Sepsis; Neonate
MeSH Terms: conditions — Sepsis | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Mechanically ventilated neonates will receive the usual protocol of sepsis and a placebo without vitamin C.
  Interventions: Drug: Placebo
- Vitamin C group (Experimental): Mechanically ventilated neonates will receive the usual protocol of sepsis plus vitamin C with a loading dose of 0.5 gm /kg and a maintenance dose of 0.5 gm /kg/hour adjusted for six hours for 7-10 days.
  Interventions: Drug: Vitamin C

INTERVENTIONS:
Drug: Placebo — Mechanically ventilated neonates will receive the usual protocol of sepsis and a placebo without vitamin C.
  Arms: Control group
Drug: Vitamin C — Mechanically ventilated neonates will receive the usual protocol of sepsis plus vitamin C with a loading dose of 0.5 gm /kg and a maintenance dose of 0.5 gm /kg/hour adjusted for six hours for 7-10 days.
  Arms: Vitamin C group

SUMMARY:
This study aims to evaluate the effect of intravenous vitamin C infusion on septic mechanically ventilated full-term neonates who underwent surgical interventions regarding mechanical ventilation parameters, time to wean, and the need for inotropic support.

DETAILED DESCRIPTION:
Neonatal sepsis is a syndrome featuring non-specific signs and symptoms of systemic infection accompanied by bacteremia in the first 28 days of extrauterine life. This condition is a public health problem that still contributes to mortality and morbidity in neonatal intensive care units (NICUs) in high, as well as low- and middle-income countries.

Vitamins are essential micronutrients with key roles in many biological pathways relevant to sepsis. Some of these relevant biological mechanisms include antioxidant and anti-inflammatory effects, protein and hormone synthesis, energy generation, and regulation of gene transcription.

Vitamin C, ascorbic acid, is a water-soluble essential micronutrient commonly found in plants, especially fruits. When absorbed, it dissociates at physiological pH to form ascorbate, the redox state of the vitamin most commonly found in cells. In addition to being a potent antioxidant, vitamin C is a cofactor for enzymes involved in protein and hormone synthesis, metabolic pathways for energy generation, and regulation of gene transcription.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 37 weeks.
* Both sexes.
* Neonates with sepsis are diagnosed both clinically and serologically after any surgical intervention.

Exclusion Criteria:

* Major congenital anomalies and Chromosomal abnormalities.
* neonate <37weeks gestation.
* Hypoxic Ischemic Encephalopathy (HIE).
* Neuromuscular diseases.
* Intraventricular hemorrhage (IV Hge).

Min Age: 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Duration of mechanical ventilation | 28 days from the start of ventilation
  Duration of mechanical ventilation was recorded from start of ventilation till weaning or death.

SECONDARY OUTCOMES:
Need for inotropic support | 28 days from the start of ventilation
  Need for inotropic support was recorded.
Mortality | 28 days from the start of ventilation
  Mortality was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.

REFERENCES:
- [Derived] Elmesiry AM, Elsheikh MR, Elshimy KM, Abotaleb AM. Role of vitamin C infusion in postoperative mechanically ventilated neonates with sepsis: a randomized controlled trial. Eur J Pediatr. 2025 Nov 29;184(12):806. doi: 10.1007/s00431-025-06625-4. PMID 41315087